CLINICAL TRIAL: NCT02530814
Title: Organochlorine Pesticide Exposure in Residents Near Lake Apopka
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201401073
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Pesticide Exposure
Keywords: organochlorine compounds; pesticides
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for analysis of organochlorine pesticides and auto-antibodies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Lake Apopka Farmworkers: This group will have a onetime blood collection and questionnaires regarding health status and health concerns.
  Interventions: Other: Blood Collection
- Existing Data Group: The investigators will collect existing data from the National Health and Nutrition Examination Survey (NHANES) for the range of concentrations of these chemicals in the blood of Americans.

INTERVENTIONS:
Other: Blood Collection — Onetime blood collection.
  Groups: Lake Apopka Farmworkers

SUMMARY:
In the Lake Apopka, Florida area for over 50 years starting in the 1940s, organochlorine pesticides (OCPs) including 4,4'-dichlorodiphenyltrichloroethane (DDT), dieldrin, chlordane, toxaphene and more recently methoxychlor were sprayed on farmlands in order to control pests and to improve crop harvests. For most of those years, the farmworkers were exposed to the pesticides as part of their work. Because of their lipophilic (fat soluble) nature, these organochlorine pesticides (OCPs) are readily taken up into the body and not readily eliminated. Therefore, they can be detected in exposed individuals for many years after the exposure. There is some evidence that certain OCPs can cause or exacerbate medical problems in sensitive individuals. For example, exposure to some OCPs has been associated with development of Parkinsonism. Exposure to other OCPs has been associated with development of lupus erythematosus, an auto-immune disease. Other adverse effects of exposure to OCPs are endocrine disruption because some OCPs mimic estrogens and others mimic androgens, or may have mixed interactions with steroid receptors.

In this research study the investigators aim is to test the blood from former farmworkers during the 1940s through the late 1970s who reside in the Lake Apopka area for OCPs and for the auto-antibodies. In addition, questionnaires will provide insight on their health status and health concerns.

DETAILED DESCRIPTION:
In this research study, a onetime blood test will be collected from former farmworkers during the 1940s through the late 1970s who reside in the Lake Apopka area for OCPs and for the auto-antibodies. In addition, questionnaires will provide insight on their health status and health concerns.

The investigators will collect existing data from the National Health and Nutrition Examination Survey (NHANES) which has monitored the pesticide exposure (with the exception of toxaphene) of people older than 8 years, so there is information on the range of concentrations of these chemicals in the blood of Americans. This data will be use as the control group for comparison with the values found for OCP concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Persons who worked on farms near lake Apopka, Florida up to 1998.
* Preference will be given to those who worked on the farms for over 10 years.

Exclusion Criteria:

* Persons who did not work on farms near Lake Apopka, Florida up to 1998.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited from the Florida Farmworker Association of Florida, Lake Apopka, FL.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Blood levels of organochlorine pesticides will be compared between the groups | Day 1
  Blood collected will be analyzed for DDT, dieldrin, chlordane, methoxychlor and the metabolites of DDT and methoxychlor. The data will be compared between the groups.

SECONDARY OUTCOMES:
Level of auto-antibodies will be recorded | Day 1
  Blood collected will be analyzed for measurement of auto-antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Margaret O. James, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Age and years worked on farms will be shared
Supporting Information: Study Protocol, ICF
Time Frame: Will be reported in publication, in preparation.
Access Criteria: upon request

REFERENCES:
- [Background] Beard J; Australian Rural Health Research Collaboration. DDT and human health. Sci Total Environ. 2006 Feb 15;355(1-3):78-89. doi: 10.1016/j.scitotenv.2005.02.022. PMID 15894351
- [Background] Eskenazi B, Chevrier J, Rosas LG, Anderson HA, Bornman MS, Bouwman H, Chen A, Cohn BA, de Jager C, Henshel DS, Leipzig F, Leipzig JS, Lorenz EC, Snedeker SM, Stapleton D. The Pine River statement: human health consequences of DDT use. Environ Health Perspect. 2009 Sep;117(9):1359-67. doi: 10.1289/ehp.11748. Epub 2009 May 4. PMID 19750098
- [Background] Xu X, Dailey AB, Talbott EO, Ilacqua VA, Kearney G, Asal NR. Associations of serum concentrations of organochlorine pesticides with breast cancer and prostate cancer in U.S. adults. Environ Health Perspect. 2010 Jan;118(1):60-6. doi: 10.1289/ehp.0900919. PMID 20056587
- [Background] Chhillar N, Singh NK, Banerjee BD, Bala K, Mustafa M, Sharma D, Chhillar M. Organochlorine pesticide levels and risk of Parkinson's disease in north Indian population. ISRN Neurol. 2013 Jul 8;2013:371034. doi: 10.1155/2013/371034. Print 2013. PMID 23936670
- [Background] Wang F, Roberts SM, Butfiloski EJ, Morel L, Sobel ES. Acceleration of autoimmunity by organochlorine pesticides: a comparison of splenic B-cell effects of chlordecone and estradiol in (NZBxNZW)F1 mice. Toxicol Sci. 2007 Sep;99(1):141-52. doi: 10.1093/toxsci/kfm137. Epub 2007 Jun 19. PMID 17578864